CLINICAL TRIAL: NCT02604784
Title: Feasibility, Efficacy and Safety of Pressurized IntraPeritoneal Air-flow Chemotherapy (PIPAC) With Oxaliplatin, Cisplatin and Doxorubicin in Patients With Peritoneal Carcinomatosis From Colorectal, Ovarian, Gastric Cancers and Primary Tumors of the Peritoneum: An Open-label, Two-arms, Phase I-II Clinical Trial. PI-CaP
Brief Title: Study of Efficacy and Safety of Laparoscopic Intra-abdominal Chemotherapy (PIPAC) Performed in Patients With Peritoneal Carcinomatosis From Colorectal, Ovarian, Gastric Cancer and Primary Peritoneal Tumors
Acronym: PI-CaP
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Fondazione del Piemonte per l'Oncologia (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 015-IRCCS-27F-1
Record Dates: First submitted 2015-11-03; First posted 2015-11-13 (Estimated); Last update posted 2020-09-17 (Actual); Status verified 2020-09

CONDITIONS: Peritoneal Carcinomatosis
Keywords: Pressurized Intra Peritoneal Air-flow Chemotherapy (PIPAC); Chemotherapy; Peritoneal Carcinomatosis
MeSH Terms: conditions — Peritoneal Neoplasms | interventions — Cisplatin; Doxorubicin; Oxaliplatin

STUDY DESIGN:
Intervention Model Description: Two parallel cohorts according to patients characteristics Patient with indication for systemic standard chemotherapy will be accrued in Cohort A (for a Phase II repeated single dose PIPAC).
  Patient with no indication for sistemic standard chemotheralpy will be accrued in Cohort B ( for a Phase, single ascending dose PIPAC)
Oversight: Data Monitoring Committee: No

ARMS (2):
- cohort A (Experimental): Cohort A: For patients that have indication for systemic therapy with standard chemotherapy. This cohort has a phase II design; the Objective Response Rate (ORR) will be evaluated according to the RECIST criteria (version 1.1) after 2 and 3 cycles of PIPAC with Cisplatin (7.5 mg/m²) + Doxorubicin (1.5 mg/m2 ) or Oxaliplatin (92 mg/m2) according to the primary cancer, in association with standard systemic chemotherapy.
  Interventions: Drug: Pressurized IntraPeritoneal Air-flow Chemotherapy (PIPAC) fixed repeated dose
- cohort B (Experimental): Cohort B: For patients that have not indication for systemic therapy with standard chemotherapy. This cohort has a phase I design; with a dose-escalation design the maximum tolerated doses and recommended doses of Cisplatin + Doxorubicin and Oxaliplatin (according to the pathology) administered through PIPAC in patients with peritoneal carcinomatosis will be evaluated.
  Interventions: Drug: Pressurized IntraPeritoneal Air-flow Chemotherapy (PIPAC) increasing single dose

INTERVENTIONS:
Drug: Pressurized IntraPeritoneal Air-flow Chemotherapy (PIPAC) fixed repeated dose — An open access with a midline 5-6 cm incision is performed and a single-port platform is positioned. A 12 mm Hg CO2 pneumoperitoneum is inflated. PC extent is evaluated according to Peritoneal Cancer Index (PCI) and peritoneal biopsies are taken. A nebulizer is connected to an intravenous high-pressure injector and inserted into the peritoneal cavity; the tightness of the abdomen has to be documented with a CO2 zero-flow. The laparoscopic camera and the nebulizer are maintained in position by a self-retaining retractor (Thompson). A pressurized aerosol containing drugs is delivered. Standard dosage of drugs for each PIPAC: Cisplatin (7.5 mg/m²) + Doxorubicin (1.5 mg/m²) or Oxaliplatin (92 mg/m²) The capnoperitoneum is then maintained for 30 minutes at 37°C. At the end, the aerosol is exsufflated through two sequential micro-particle filters into the air-waste system of the hospital.
  Other Names: Cisplatin + Doxorubicin in ovarian, gastric cancer and in primary peritoneal tumors; or Oxaliplatin in colorectal cancer
  Arms: cohort A
Drug: Pressurized IntraPeritoneal Air-flow Chemotherapy (PIPAC) increasing single dose — An open access with a midline 5-6 cm incision is performed and a single-port platform is positioned. A 12 mm Hg CO2 pneumoperitoneum is inflated. PC extent is evaluated according to Peritoneal Cancer Index (PCI) and peritoneal biopsies are taken. A nebulizer is connected to an intravenous high-pressure injector and inserted into the peritoneal cavity; the tightness of the abdomen has to be documented with a CO2 zero-flow. The laparoscopic camera and the nebulizer are maintained in position by a self-retaining retractor (Thompson). A pressurized aerosol containing drugs is delivered. Escalating dosage of drugs for PIPAC: Cisplatin + Doxorubicin (from 15 mg/m² + 3 mg/m² to 100 mg/m² + 30 mg/m²) or Oxaliplatin (from 92 mg/m² to 300mg/m²).The capnoperitoneum is then maintained for 30 minutes at 37°C. At the end, the aerosol is exsufflated through two sequential micro-particle filters.
  Other Names: Cisplatin + Doxorubicin in ovarian, gastric cancer and in primary peritoneal tumors; or Oxaliplatin in colorectal cancer
  Arms: cohort B

SUMMARY:
Single center, open label, phase I-II, non-randomized, two-cohort, repeated single dose study to explore the feasibility, efficacy, safety, and Overall Response Rate (ORR) of oxaliplatin, or cisplatin and doxorubicin when given as a pressurized intraperitoneal chemotherapy (PIPAC) to patients (men and women) with peritoneal carcinomatosis from ovarian, gastric and colorectal cancers and in primary cancers of peritoneum.

ELIGIBILITY:
Inclusion Criteria:

* Clinical and pathological confirmation of peritoneal carcinomatosis from gastric, colorectal and ovarian cancers or primary peritoneal tumors.
* Patients aged between 18 and 78 years.
* Performance status sec. ECOG ≤ 2
* Disease progression/relapse after at least one line of previous i.v. standard chemotherapy in gastric cancer and primary peritoneal tumors and two lines in colorectal and ovarian cancers.
* Patients with peritoneal carcinomatosis from ovarian, gastric and colorectal cancers and primary peritoneal cancers not eligible to cytoreductive surgery +/- HIPEC.
* Blood and electrolyte counts, liver, renal and cardiopulmonary function parameters within 10% of the normal range.
* Written informed consent.
* Tumor mass present on CT-scan in order to allow tumor response assessment with RECIST-criteria.

Exclusion Criteria:

* Extra-abdominal metastatic disease, with the exception of isolated pleural carcinomatosis.
* Bowel obstruction.
* Severe renal impairment, myelosuppression, severe hepatic impairment, severe myocardial insufficiency, recent myocardial infarction, severe arrhythmias.
* Immunocompromised patients such as those with an immunosuppressive medication or a known disease of the immune system.
* Creatinine clearance < 60 ml /min.
* Pregnancy.
* Previous treatment reaching the maximum cumulative dose of doxorubicin, daunorubicin, epirubicin, idarubicin and/or other anthracyclines and anthracenediones.
* Known allergy to cisplatin or other platinum-containing compounds or to doxorubicin.
* Patients of both sexes who do not conduct complete abstinence from heterosexual relationships or agree to use an effective clinically acceptable method (with failure rate <1%) during the study and the following 6 months after the last treatment.

Ages: 18 Years to 78 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2015-10; Primary Completion 2020-05-31 (Actual); Study Completion 2020-05-31 (Actual)

PRIMARY OUTCOMES:
Overall Response Rate (ORR) according to RECIST criteria (version 1.1) after 2 and 3 cycles of PIPAC. | 18 weeks

SECONDARY OUTCOMES:
The overall survival (OS) | 30 months
The degree of histological regression assessed by pathological review | 18 weeks
The median time to progression (TTP) according to RECIST criteria (version 1.1) after two or three cycles of PIPAC | 30 months
Measurement of clinical tumor response to therapy using FDG- Positron Emission Tomography (PET) according to PERCIST criteria (version 1.0). | 22 weeks
The Peritoneal Carcinomatosis Index (PCI) before and after therapy | 18 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Surgical Oncology - FPO-IRCCS Institute for Cancer Research and Treatment, Candiolo, Turin, Italy

REFERENCES:
- [Derived] Robella M, Berchialla P, Borsano A, Cinquegrana A, Ilari Civit A, De Simone M, Vaira M. Study Protocol: Phase I Dose Escalation Study of Oxaliplatin, Cisplatin and Doxorubicin Applied as PIPAC in Patients with Peritoneal Metastases. Int J Environ Res Public Health. 2021 May 25;18(11):5656. doi: 10.3390/ijerph18115656. PMID 34070561